CLINICAL TRIAL: NCT02151695
Title: Phase 2 Study of Safety and Efficacy of Aflibercept in Proliferative Diabetic Retinopathy.
Brief Title: Safety and Efficacy of Aflibercept in Proliferative Diabetic Retinopathy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: mEdICARE
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2019-03

CONDITIONS: Naive Patients With Uncomplicated Proliferative Diabetic Retinopathy

ARMS (2):
- Panretinal photocoagulation (Active Comparator)
  Interventions: Procedure: panretinal photocoagulation
- Aflibercept intravitreal injections (Experimental)
  Interventions: Drug: Aflibercept intravitreal injections

INTERVENTIONS:
Procedure: panretinal photocoagulation
  Arms: Panretinal photocoagulation
Drug: Aflibercept intravitreal injections
  Arms: Aflibercept intravitreal injections

SUMMARY:
Proliferative diabetic retinopathy is a serious complication of diabetes mellitus, partly consecutive to upregulation of vascular endothelial growth factor (VEGF) as a consequence of retinal ischemia leads. Aflibercept has been approved by FDA and European medicine agency for treatment of exudative age-related macular degeneration, another retinal disease characterized by choroidal new vessels.

The aim of this pilot study is to evaluate the efficacy and the safety of Aflibercept intravitreal injections compared to panretinal photocoagulation for proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus type 1 or type 2 complicated by PDR
* Male or female over 18 years
* HbA1c <11.6% at study entry
* Systolic blood pressure <160 mmHg and diastolic blood pressure <105 mmHg at study entry
* Backgrounds clear eye, pupil dilation and patient cooperation sufficient to allow examination or fundus photographs of good quality

Exclusion Criteria:

* Hypersensitivity to aflibercept or to any of the excipients
* History of retinal laser (macular or panretinal photocoagulation), of intravitreal injections, of vitrectomy in the eye studied
* PDR associated with tractional retinal detachment in the eye studied
* PDR associated with fibrovascular proliferation in the eye studied
* Florid diabetic retinopathy
* Eye infection or periocular active or suspected
* Unbalanced glaucoma in the eye studied
* Other eye disease in the eye studied
* Patients with significant medical problems that may interfere with the evaluation of the safety or efficacy of the treatment studied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with regression of retinal neovascularization between baseline and 12th month. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEVEZIEL, MD, PhD, Principal Investigator — Poitiers University Hospital
Locations (1):
- Chu de Poitiers, Poitiers, France